CLINICAL TRIAL: NCT03276494
Title: Intraosseous Administration of Hypertonic Saline in Acute Brain-injured Patients: A Prospective Case Series and Literature Review
Brief Title: Safety & Tolerability of Hypertonic Saline Administration Via Intraosseous Access
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Archana Hinduja, Assistant Professor Division of Cerebrovascular Disease and Neurocritical Care, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017H0067
Record Dates: First submitted 2017-06-29; First posted 2017-09-08 (Actual); Results first posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-06

CONDITIONS: Stroke; Intracranial Hypotension; Cerebral Edema
MeSH Terms: conditions — Stroke; Intracranial Hypotension; Brain Edema | interventions — Saline Solution, Hypertonic

STUDY DESIGN:
Intervention Model Description: prospective case series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Intraosseous (Other): Administration of intraosseous hypertonic saline
  Interventions: Device: Intraosseous; Drug: Hypertonic saline

INTERVENTIONS:
Device: Intraosseous — Intraosseous administration of hypertonic saline
Drug: Hypertonic saline — Intraosseous administration of hypertonic saline

SUMMARY:
Hypertonic saline is used to treat elevated intracranial pressure. Intraosseous vascular access has been used to administer fluids and medications. This study combines these to administer 3% hypertonic saline via IO.

DETAILED DESCRIPTION:
HTS is used to mitigate and temporize intracranial pressure (ICP) elevations and cerebral edema by creating an osmotic gradient across the cell wall. HTS is part of the elevated ICP algorithm in the emergency neurologic life support protocols HTS is superior to mannitol which is the alternate osmotherapy agent . HTS is typically administered via central vascular access due to the concern that if extravasation of the infusion occurs, tissue damage from cell implosion can occur

The IO route is generally accepted in resuscitation environments including the emergency department, EMS, and military settings with some authors recommending the IO as a primary method of obtaining emergency vascular access The adult advanced cardiac life support (ACLS) guidelines recommend either intravenous or IO access.

A number of studies have established the safety of IO administration of hypertonic solutions. Randomized adult pigs to IO 7.5% HTS, IO 3% HTS, and 0.9% isotonic saline and found regular tissue morphology, no necrosis or microscopic ischemic changes in the HTS groups. Several studies conducted to evaluate the efficacy of hypertonic solutions on resuscitation for hemorrhagic shock used the IO route and did not make note of problems arising from the administration of IO HTS. Another study using a canine model of hemorrhagic shock briefly mentioned transient lameness in the IO HTS group, but this resolved by 48 hours . While the majority of studies using hypertonic saline solutions did not make note of complications, one study induced hemorrhagic shock in dehydrated swine and resuscitated one group with 7.5% HTS and noted a high rate of local complications from soft tissue and bone marrow necrosis .

One study noted a subgroup of patients in which IO access was obtained on conscious patients. None of the patients received local anesthetic and none reported pain during insertion. Eighteen of the 22 conscious patients reported pain during fluid administration. Central venous catheter (CVC) placement is the current standard of care; even with local anesthesia it can be painful. Most of the potential subjects, due to the nature of their severe neurologic injury, may not be affected by the pain associated with IO fluid administration. Manufacturer literature suggests the use of lidocaine to anesthetize the bone before infusing if possible (Teleflex).

It is expected that utilizing IO for vascular access in the ICU will be safe and tolerable. If this study confirms the anticipated results, there are numerous implications. First, neurologically injured patients requiring emergent HTS may have faster access to this therapy. A study comparing IO to CVC access undergoing resuscitation in the emergency department found IO to be faster to insert (2.3 vs. 9.9 minutes) and had fewer failures to access on the first attempt. Second, serious complications from IO were absent compared with severe to life-threatening mechanical complications from CVC including pneumothorax, damage to the carotid artery, and bleeding which were cited at 0.7%-2.1% depending on site. And thirdly, central line associated blood stream infections (CLABSI) are a leading cause of hospital acquired infections in the ICU and are associated with higher mortality. CLABSI rates are measured by number of infections per 1,000 catheter days and shorter CVC dwell time is prudent. If a reliable and rapid source of vascular access could postpone or eliminate CVC insertion, risk of CLABSI may be reduced. These potential benefits outweigh the minimal expected risk.

ELIGIBILITY:
Inclusion Criteria:

* NCCU patients in which osmotherapy with HTS is planned (standard of care
* Does not already have a CVC or PICC.

Exclusion Criteria:

* <18 years old
* Known pregnancy
* Long bone fracture in the targeted site
* Proximity to prosthetic joint
* Excessive tissue/absence of anatomical landmarks
* History of osteopetrosis
* Previous significant orthopedic procedure at site
* Prosthetic limb or joint
* IO catheter use in the past 48 hours of the target bone
* Infection at the area of insertion
* Hypersensitivity to lidocaine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2018-04-21 (Actual); Study Completion 2018-04-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
manuscript on the case series has been submitted
Supporting Information: CSR

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intraosseous
Started | 6
Completed | 5
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intraosseous
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 2
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Tissue Damage
Description: Number of subjects with tissue damage (e.g. Myonecrosis, Skin necrosis, Extravasation, Compartment syndrome, Osteomyelitis). These data points will be determined by clinician assessment.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Intraosseous
Number analyzed (Participants) | 5
Participants | 0

2. Secondary Outcome: Pain Scale
Description: Pain (CPOT-critical care pain observation tool). All non-verbal subjects have pain assessed with a CPOT score, as observed by clinicians. The CPOT is a validated pain score for nonverbal patients. This tool assesses pain with nonverbal indicators, adding 1-2 points for several nonverbal indicators of pain, 0 if the nonverbal indicator is absent, and is reported as a total summed score. It ranges from 0-8, with 0 indicating no pain and 8 indicating high pain.
  No patients were verbal, so the numeric pain rating scale was not used for any patients.
Time Frame: 24 hours
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Intraosseous
Number analyzed (Participants) | 5
units on a scale | 0 [0 to 6]

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Intraosseous
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/94/NCT03276494/Prot_000.pdf